CLINICAL TRIAL: NCT05268991
Title: Aging Biomarkers, Geriatric Assessment and Electronic Frailty Index (AGE)
Brief Title: Aging and Frailty Study
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00080711; WFBCCC 04721 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2022-02-15; First posted 2022-03-07 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Effects of Chemotherapy; Aging; Frailty
MeSH Terms: conditions — Frailty | interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AGE Participants: Participants aged 65 and older with diagnosis of solid tumor malignancy or lymphoma and planned to start a new chemotherapy regimen in the outpatient setting
  Interventions: Other: Geriatric Assessments and Frailty Indices

INTERVENTIONS:
Other: Geriatric Assessments and Frailty Indices — Eligible and consented subjects will undergo a baseline assessment prior to chemotherapy initiation inclusive of geriatric/frailty assessments, patient reported outcomes and blood samples for biomarkers of aging. Assessment measures and blood samples will be repeated post cycle 1 and 2 of chemotherapy. Toxicity will be recorded from the medical record

SUMMARY:
The purpose of this research study is to compare methods to help personalize the prediction of chemotherapy side effects for older adults and to evaluate whether chemotherapy causes changes in the body that are associated with aging.

DETAILED DESCRIPTION:
Primary Objective: Describe mean and variation of the electronic frailty index-cancer, geriatric measures, patient reported outcomes, and biomarkers of aging of chemotherapy, and their change.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and older
* Planned to initiate a new chemotherapy regimen
* Solid tumor malignancy of any stage or lymphoma
* Any performance status
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).
* Life expectancy of ≥3 months

Exclusion Criteria:

* Initiating biologic, endocrine or immunotherapy only.
* Hematologic malignancy other than lymphoma.
* Concurrent radiation therapy.
* Planned inpatient chemotherapy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Eligible participants will be identified by oncology providers, EPIC reports, or through screening of clinic schedules by the Cancer Control Survivorship Disease Oriented Team Clinical Trial Coordinator or research nurse
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Resiliency Administered Assessments - Change of Short Physical Performance Battery (SPPB) | At baseline, 3 months and 6 months after chemotherapy
  The SPPB will be used to assess lower extremity physical function (a short walk of 4 meters, timed repeated chair stands and balances tests). Each task is scored ranging from 0-4 (0 = unable to complete; 4 = highest performance level) with the total sum score range from 0-12. Lower scores indicate increased risk of disability, hospitalization and worse survival among older adults with and without cancer.
Resiliency Administered Assessments - Change of Grip Strength | At baseline, 3 months and 6 months after chemotherapy
  Grip strength in both hands will be measured using an adjustable, hydraulic grip strength dynamometer. Two trials will be conducted for each hand. Frailty by this criterion is defined by grip strength cutoffs which are dependent upon both gender and body mass index.
Resiliency Administered Assessments - Change of Blessed Orientation Memory and Concentration Test (BOMC) | At baseline, 3 months and 6 months after chemotherapy
  A 6 item test that provides a measure of cognition. For items to 1 to 3 the response is either correct (score = 0) or incorrect (score = 1). For items 4 to 6, one point is added for each error (items 4 and 5 maximum error = 2; item 6 maximum error = 5). Maximum score = 28. Participants with scores ≥ 11 will receive further evaluation or intervention as deemed medically appropriate by the treating physician.
Change of Electronic Frailty Index and Cancer Score/Category | At baseline, 3 months and 6 months after chemotherapy
  Measures collected from the resiliency assessments (Short Physical Performance Battery, Grip Strength, Blessed Orientation Memory and Concentration Test) will be used to calculate the Fried Frailty Index (FFI) to assess frailty. Scores will be anchored to the date of each assessment time point (i.e., baseline visit, follow-up visits). Each data element will be scored from 0 to 1 and the mean will be computed to calculate the overall score. Some data elements (e.g., comorbidities) will be coded as absent or present (0 or 1) and some (e.g., body mass index) will be assigned a score that ranges from 0 to 1. The higher score indicates a higher frailty of the participant.
Change in Patient Reported Outcomes Measurement - PROMIS 29 | At baseline, 3 months and 6 months after chemotherapy
  Measures collected from this is a 29-item self-reported measure including 4 items each for the following domains: physical function, anxiety, depression, fatigue, sleep disturbance, social function, and pain interference; plus 1 item measuring average pain intensity and cognition. Scoring is based on a 1-5 point Likert scale (1 = very often; 5 = never). Items are summed to create a total score that ranges from 6-30 and lower scores indicate greater self-reported difficulty.
Change of Biomarkers of Aging Observed During Study Intervention | At baseline, 3 months and 6 months after chemotherapy
  Investigators will measure targeted panels of blood-based biomarkers including but not limited to serum Interleukin-6, tumor necrosis factor receptors, growth differentiating factor 15, and cystatin C.
Number of Incidences of Toxicity - Grades 2 to 5 Related to Standard of Care Chemotherapy | Up to 6 months after chemotherapy
  Grade 2 to 5 incidences of toxicities will be recorded and measured using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Number of Documented Dose Reductions During Chemotherapy | Up to 6 months after chemotherapy
  Participants that have the chemotherapy doses reduced during treatment will be documented.
Number of Dose Delays During Chemotherapy | Up to 6 months after chemotherapy
  Dose delays greater than three days from planned treatment will be documented.
Number of Early Discontinuations of Chemotherapy | Up to 6 months after chemotherapy
  Participants that have chemotherapy discontinued prior to anticipated completion of treatment will be documented.
Number of Unplanned Hospitalizations | Up to 6 months after chemotherapy
  Participants that required unplanned hospitalizations will be documented.
Overall Survival | Up to 6 months after chemotherapy
  Participants will be followed after completion of chemotherapy for survival status.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Klepin, MD, MS, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No